CLINICAL TRIAL: NCT04309201
Title: Relationship With Muscle Wasting and Insulin Resistance in a Group of Non-diabetic Hemodialysis Patients.
Brief Title: Insulin Resistance, Sarcopenia and Plasma BAIBA Levels
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 108084
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Sarcopenia; Insulin Resistance
Keywords: Insulin resistance; Sarcopenia; β-aminoisobutyric acid
MeSH Terms: conditions — Sarcopenia; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Insulin resistance (IR) is an early metabolic alteration in chronic kidney disease (CKD) patients, becoming almost universal in those who reach the end stage of kidney failure. The skeletal muscle represents the primary site of IR in CKD, and alterations at sites beyond the insulin receptor are recognized as the main defect underlying IR in this condition. The etiology of IR in CKD is multifactorial in nature and may be secondary to disturbances that are prominent in renal diseases, including physical inactivity, chronic inflammation, oxidative stress, vitamin D deficiency, metabolic acidosis, anemia, adipokine derangement, and altered gut microbiome.

IR has been solidly associated with intermediate mechanisms leading to cardiovascular (CV) disease in CKD including left ventricular hypertrophy, vascular dysfunction, and atherosclerosis. Recent studies have identified a muscle factor β-aminoisobutyric acid (BAIBA), which is produced by skeletal muscle during physical activity. BAIBA have been found to link with sedentary life style, abdominal obesity, and impairments in carbohydrate and lipid metabolism. A few studies have shown that BAIBA can protect from diet-induced obesity in animal models. It induces transition of white adipose tissue to a "beige" phenotype, which induces fatty acids oxidation and increases insulin sensitivity. While the exact mechanisms of BAIBA-induced metabolic effects are still not well understood, the aim of this study is want to study its relationship with muscle wasting and insulin resistance in a group of non-diabetic hemodialysis patients.

DETAILED DESCRIPTION:
Study Design and Population

Patients and Methods

This study is an observational, cross-sectional and prospective cohort study. One hundred and fifty patients on non-diabetic hemodialysed patients will be included for the cross-sectional survey; Twenty healthy subjects will be elected as the controls. Prevalent adult HD patients with dialysis vintages over 3 months will be recruited. Patients are maintained on regular HD prescription, three times a week, for four-hour sessions. Subjects with significant comorbid conditions such as cancer, heart failure, or severe liver disease and chronic infection such diabetic foot will be excluded. This study is conducted according to the guidelines laid down in the Declaration of Helsinki, and all procedures were reviewed as well as approved by the Regional Hospital Ethics Committee. All subjects should give their written informed consent to participate in the study. Subjects' demographic and clinical characteristics, including age, gender, weight, height, body mass index (BMI), dialysis vintage, and Kt/V will be recorded, and comorbidities and current therapies will be collected.

Anthropometric and biochemical assessments

Systolic and diastolic blood pressures are taken with the subjects in the supine position. A measurement of height and weight was performed on all subjects. Waist circumference was measured at the midpoint between the lower border of the rib cage and the iliac bone. The concentration of plasma insulin was assayed by radioimmunoassay. Fasting plasma glucose was measured using the glucose oxidase method. HbA1c was measured by affinity chromatography. Total cholesterol, triglyceride, and HDL cholesterol levels were measured enzymatically using an autoanalyzer (Hitachi 747; Hitachi, Tokyo, Japan). Serum insulin concentrations are determined by IRMA. Adiponectin and leptin concentrations are measured using a commercially available ELISA kit.

Sample preparation

In each subject, the blood samples are drawn from the arteriovenous fistula in of each participant in the morning after fasting for at least 8 h and on the day of hemodialysis. The samples are properly processed, refrigerated at 2-8 C, and the plasma is separated immediately by centrifugation. Each serum sample is heat-inactivated by incubation at 65 C for 30 min. Fetal bovine serum (FBS; Gibco BRL, Grand Island, NY, USA), a negative control, is treated with activated charcoal (Sigma, St. Louis, MO, USA) overnight at 4 C and filtered to remove all small molecules and AhR agonists that might have been present. TCDD, a positive control for AhR agonists, was purchased from Sigma Co. Plasma BAIBA levels are assessed by a Liquid chromatography-tandem mass spectrometry (LC-MS/MS) method, as previously described (15). Cell-based AhR ligand activity (CALA) assay and ELISA assay will be performed (16)

HOMA-IR, HOMA-%B, HOMA-%S, and disposition index are calculated by the following formulae.

HOMA-IR1 = [fasting insulin (mU/l) × fasting glucose(mg/dl)× 0.0555]/22.5 HOMA-%B1 = [20 × fasting insulin (mU/l)]/[(fasting glucose(mg/dl) × 0.0555)-3.5] HOMA-%S1 = [1/ HOMA-IR1] × 100% Disposition index 1= (HOMA-%S1/100) × (HOMA-%B1/100)

Dual-Energy X-ray Absorptiometry (DEXA)

DEXA is a widely used reference method for body FFM and FM measurements.(10) DEXA was performed using a Lunar Prodigy (GE Medical Systems, Madison, WI). Whole-body scans were performed according to manufacturer's instructions, and body FM (FMDEXA), LTM (LTMDEXA) and bone mineral content were analyzed using the manufacturer's software. The DEXA method uses an X-ray tube with a filter to generate low-energy (40 kV) and high-energy (70 or 100 kV) photons. When photons at different energy levels pass through tissue, their absorptions can be expressed as a ratio of attenuation at lower or higher energy levels. DEXA estimate of FFM was calculated as a sum of LTMand bone mineral content estimates. All patients were examined by the same observer.

Bioelectric Impedance Spectroscopy

Whole-body bioelectric impedance spectroscopy (BIS) measurement using a body composition monitor (BCM: Fresenius Medical Care, Bad Homburg, Germany) was performed on each of the participants enrolled in the study by a specific member of the staff who had completed a training course in the BCM technique. The BCM measures the impedance spectroscopy at 50 different frequencies between 5 kHz and 1 MHz. Measurements were taken on the day before dialysis with the patient calm, supine, and relaxed in the dialysis bed for 10minutes. Four electrodes were placed on the patient's hand and foot on the side contra lateral to their arteriovenous fistula. Specific exclusion criteria were dictated by the device and included history of a pacemaker, defibrillator, metallic sutures, or stent implantation and amputation of a major limb. As a multifrequency bioimpedance device, BCM not only provides extracellular (ECWBCM), intracellular (ICWBCM), and total body water (TBWBCM) measurements but also estimates the body composition in terms of lean tissue mass (LTMBCM-mainly muscle), fat mass (FATBCM), adipose tissue mass (ATMBCM-mainly fat), and overhydration (OH) according to the body compositionmodel.(17) This device combined BIS with the BCM model described in Chamney et al,11 and it takes into account the dissimilar hydration of relevant tissues. Briefly, the device was modified to reflect the presence of excess fluid accumulated due to pathologic reasons, that is, patients with kidney failure. It has therefore set constants for each of the body composition compartment. This device has been shown to be as precise as the gold standardreference methods and has been validated against reference methods for volume status and body composition assessments in healthy and HD populations, with methods frequently used in the 4-compartment model. The percentage proportions of LTMBCM, FATBCM, andATMBCM were denoted accordingly as pLTMBCM, pFATBCM, and pATMBCM.

Muscle Strength

The muscle function will be assessed on the same day of the recruitment immediately before starting the HD session by handgrip strength measurement, using a handle dynamometer. The test is performed conducting three attempts with each hand, and the mean of the strongest hand is used to determine muscle strength

ELIGIBILITY:
Inclusion Criteria:

* Received stable hemodialysis at least 3 months

Exclusion Criteria:

* cancer
* heart failure
* severe liver disease
* chronic infection such diabetic foot

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hemodialysis (HD) patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Analysis of biomarkers of β-aminoisobutyric Acid( L-BAIBA) levels | 1 years
  BAIBA can protect from diet-induced obesity in animal models. It induces transition of white adipose tissue to a "beige" phenotype, which induces fatty acids oxidation and increases insulin sensitivity.

SECONDARY OUTCOMES:
Presence of Sarcopenia | 1 years
  To evaluate the association of sacropenia defined according to 1. Muscle Strength 2. Bioelectric Impedance Spectroscopy 3. Dual-Energy X-ray Absorptiometry (DEXA)

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan